CLINICAL TRIAL: NCT03903627
Title: Effect of Verbal Instruction on Pelvic Floor Muscle Contraction in Post Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Collaborators: Ariel University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0026-18-LOE
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2019-04

CONDITIONS: Pelvic Floor Muscle Weakness
Keywords: verbal cue, pelvic diaphragm, stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: all participants will receive the same verbal instruction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Verbal instruction (Experimental): The participants will be verbal instructed to contract the pelvic floor muscle with the following sentences:
  (1) "contract your pelvic floor - all sphincters"; (2) "contract your anus"; (3) "contract your pelvic floor as if you're trying to stop urinating".
  Those who will not be able to contract will be taught by the ultrasound as a biofeedback.
  Interventions: Other: verbal instruction

INTERVENTIONS:
Other: verbal instruction — Verbal instruction for pelvic floor contraction will be given to participants. Ultrasound examination will be conducted to asses urinary bladder displacement being a marker for pelvic floor muscle function.
  Other Names: transabdominal ultrasound assesment

SUMMARY:
The aim of this study is to investigate which verbal instruction will lead to the most efficient contraction of pelvic floor muscles in post stroke patients. Pelvic floor muscle contraction will be evaluated via transabdominal ultrasound. ultrasound.

DETAILED DESCRIPTION:
Sub-acute stroke patients during the rehabilitation period in the rehabilitation hospital will be examined. Each participant will be asked to contract the pelvic floor muscles using three different verbal instructions: (1) "contract your pelvic floor - all sphincters"; (2) "contract your anus"; (3) "contract your pelvic floor as if you're trying to stop urinating". Those who will not be able to contract will be taught by the ultrasound as a biofeedback.

The assessment of pelvic floor contraction will be measured by measuring bladder displacement via abdominal ultrasound. A curved linear array transducer will be placed in the transverse plane immediately suprapubically over the lower abdomen angled at 15-30 degrees from the vertical. An on screen caliper and measurement tool will be used to measure bladder displacement.

ELIGIBILITY:
Inclusion Criteria:

* one to 6 months post first stroke
* understand the language and simple instruction
* willing to participate in the study
* mini mental assessment >21

Exclusion Criteria:

* Aphasia
* side neglect
* active urinary tract infection
* has been treated before for pelvic floor rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
urinary bladder displacement in millimeters during verbal instructions | baseline
  bladder displacement will be measured via diagnostic ultrasound using the on screen caliper tool

SECONDARY OUTCOMES:
International Consultation on Incontinence Questionnaire | baseline
  questionnaire regarding symptoms of urinary incontinence,scale range 0-21 points. higher values represent worse outcome
pelvic floor muscles endurance of contraction in seconds | baseline
  time of muscle contraction will be measured during the last contraction in each instruction
Functional Independence Measurement (FIM) tool | baseline
  assess and grade the functional status of a person based on the level of assistance he or she requires

CONTACTS AND LOCATIONS:
Overall Officials: Noa Ben-Ami, PhD, Principal Investigator — Ariel University; Gali Dar, PhD, Principal Investigator — University of Haifa
Locations (1):
- Leowenstein hospital, Department of Physical Therapy, Raanana, Israel

IPD SHARING:
Plan to Share IPD: Yes
the result of the study will be analysed. a paper will be submitted to international journal with study description including methods, examination protocol results.
Supporting Information: Study Protocol, CSR
Time Frame: one year following completion of study

REFERENCES:
- [Result] Tibaek S, Jensen R, Lindskov G, Jensen M. Can quality of life be improved by pelvic floor muscle training in women with urinary incontinence after ischemic stroke? A randomised, controlled and blinded study. Int Urogynecol J Pelvic Floor Dysfunct. 2004 Mar-Apr;15(2):117-23; discussion 123. doi: 10.1007/s00192-004-1124-1. Epub 2004 Jan 31. PMID 15014939
- [Result] Shin DC, Shin SH, Lee MM, Lee KJ, Song CH. Pelvic floor muscle training for urinary incontinence in female stroke patients: a randomized, controlled and blinded trial. Clin Rehabil. 2016 Mar;30(3):259-67. doi: 10.1177/0269215515578695. Epub 2015 Apr 10. PMID 25862769
- [Result] Ben Ami N, Dar G. What is the most effective verbal instruction for correctly contracting the pelvic floor muscles? Neurourol Urodyn. 2018 Nov;37(8):2904-2910. doi: 10.1002/nau.23810. Epub 2018 Aug 28. PMID 30152550